CLINICAL TRIAL: NCT04562207
Title: Pre-operative Carriage of Respiratory VIRUSes, and Acute Respiratory Distress Syndrome After Heart Surgery - VIRUS-ATTAC
Brief Title: Pre-operative Carriage of Respiratory VIRUSes, and Acute Respiratory Distress Syndrome After Heart Surgery
Acronym: VIRUS-ATTAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 35RC19_8869_VIRUS-ATTAC
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Heart; Surgery, Heart, Functional Disturbance as Result
Keywords: extracorporal circulation; adrs
MeSH Terms: interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Addition of a nasopharyngeal swab before surgery
  Interventions: Diagnostic Test: Screening for respiratory virus infection

INTERVENTIONS:
Diagnostic Test: Screening for respiratory virus infection — Nasopharyngeal swab for screening for respiratory virus infection before surgery

SUMMARY:
The main objective of our study is to determine whether asymptomatic influenza virus carriage is associated with an increased risk of post-operative Acute Respiratory Distress Syndrome (ARDS) after cardiac surgery. Cardiac surgery patients are particularly at risk of developing ARDS with an estimated incidence of 5-10% based on the most recent data.

DETAILED DESCRIPTION:
The primary objective of our study is to determine whether asymptomatic influenza virus carriage is associated with an increased risk of post-operative Acute Respiratory Distress Syndrome (ARDS) after cardiac surgery. Cardiac surgery patients are particularly at risk of developing ARDS, with an estimated incidence of 5-10% based on the most recent data. Acute Respiratory Distress Syndrome (ARDS) is an acute pulmonary attack of inflammatory origin. ARDS is the main cause of hypoxemic postoperative respiratory distress. Hospital mortality associated with ARDS is estimated at 35-46% depending on the degree of severity, and survivors are at increased risk of cognitive decline, depression, post-traumatic stress, or musculoskeletal weakness.

Recently, asymptomatic carriage of respiratory viruses, including the influenza virus, has been identified as a potential risk factor for respiratory complications, including ARDS, after cardiac surgery. In a monocentric observational cohort, Groeneveld et al. recently reported that performing scheduled cardiac surgery during the influenza season was associated with a significantly longer duration of postoperative mechanical ventilation and a higher incidence of postoperative ARDS compared to surgery performed outside the influenza season (OR 1.85 95%CI 1.06-3.23 p=0.03). While it is estimated that up to 77% of patients with positive influenza tests are asymptomatic in the general population, the authors hypothesized that asymptomatic viral lung carriage would act as pulmonary priming, which, in combination with other types of pulmonary attacks encountered during surgery, would predispose to the genesis of ARDS. However, Groeneveld et al. had not tested any respiratory viruses in their cohort. In addition, the relatively higher influenza vaccination rate in the Netherlands in this at-risk population (77%) suggests that other types of respiratory viruses may have contributed to the observed effect.

These data are of major interest. Indeed, in France, during the 2017-2018 epidemic season, the vaccination rate of individuals at risk was only 46%, with an estimated vaccine efficacy of only 54% in elderly patients.

The aim of this study is to determine if there is an association between asymptomatic carriage of respiratory virus, especially influenza virus, and the occurrence of post-operative complications, morbidity and mortality.

If an association between asymptomatic carriage of influenza virus, or other respiratory viruses, and the occurrence of post-operative respiratory complications, including ARDS, is confirmed, a policy of routine immunization prior to cardiac surgery or postponement of scheduled surgery in the event of a positive viral test could be a simple and inexpensive strategy to reduce these complications after cardiac surgery. Pre-emptive antiviral therapy could be discussed when neither of these strategies is possible (e.g., emergency surgery).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age ;
* Benefiting from cardiac surgery under extracorporeal circulation (ECC);
* Affiliated to a social security scheme;
* And having given free, informed and written consent

Exclusion Criteria:

* Admission for heart transplantation ;
* Admission for implantation of a left heart mechanical assist device or a total artificial heart;
* Patients with fever or flu-like symptoms during preoperative assessment (headache, myalgia, cough, nasal congestion, rhinorrhea)
* Patients participating in another clinical study that may interfere with the procedures in this study
* Persons of full age subject to legal protection (judicial protection, guardianship, trusteeship), persons deprived of their liberty, pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1256 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of ARDS within 7 days after surgery related to influenza virus infection | 7 days
  Occurrence of ARDS in population with a positive test for influenza virus within 7 days after surgery according to Berlin criteria (PMID: 22797452)

SECONDARY OUTCOMES:
Occurrence of ARDS within 7 days after surgery related to respiratory virus infection | 7 days
  Occurrence of ARDS in population with a positive test for one of 16 respiratory virus within 7 days after surgery according to Berlin criteria (PMID: 22797452)
Postoperative respiratory complications | 28 days
  Number or type of postoperative respiratory complications (according to Huzelbos et al PMID: 17047215, and French recommendations SFAR-SRLF 2017)
Morbidity | 28 days
  Number or type of postoperative non respiratory complications and data of hospitalization
Mortality | 28 days
  Number of death

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Nesseler, Md, Principal Investigator — Rennes University Hospital
Locations (5):
- France (5):
  - APHP Henri Mondor, Créteil
  - CHU Nantes, Nantes
  - APHP La Pitié-Salpétrière, Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No